CLINICAL TRIAL: NCT00529711
Title: The Efficacy of Hypertonic Lactate Solution in CABG(Coronary Artery Bypass Grafting) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innogene Kalbiotech Pte. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001/IGK-KAL/DNA/04
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Low Cardiac Output
Keywords: coronary; artery; bypass; grafting; IV; cardiac output
MeSH Terms: conditions — Cardiac Output, Low | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Hypertonic lactate
  Interventions: Drug: Hypertonic lactate
- Group 2 (Active Comparator): Ringer's lactate
  Interventions: Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hypertonic lactate — Solution given parenterally as follows:
  Intraoperative 3 ml./kg BW for 15 minutes at beginning of surgery; During surgery 1.5 ml/kg BW/hour; Second loading 1.5 ml/kg BW for 15 minutes after protamin administration; Post-operative 1 ml/kg BW/hour for 12 hours.
  Other Names: Totilac
  Arms: Group 1
Drug: Ringer's lactate — Solution given parenterally as follows:
  Intraoperative 3 ml./kg BW for 15 minutes at beginning of surgery; During surgery 1.5 ml/kg BW/hour; Second loading 1.5 ml/kg BW for 15 minutes after protamin administration; Post-operative 1 ml/kg BW/hour for 12 hours.
  Arms: Group 2

SUMMARY:
Previous clinical trials with 11.2% Hypertonic Ringer's Lactate in post-operative CABG subjects have shown an increase in several cardiac performance parameters, with lesser volume of resuscitation fluid required to reach circulation volume, as compared to Sodium Chloride.It also does not cause hyperchloremic acidosis, which is of value in treating shock patients.

The primary objectives of this prospective, randomized, open-label trial are to evaluate the clinical efficacy of hypertonic lactate in comparison to Ringer's lactate to maintain hemodynamic stability in intra- and post-CABG subjects in relation to hemodynamic status and body fluid balance, as well as to assess its safety in terms of lab parameters and occurrence of adverse events.The secondary objectives are to evaluate comparative clinical efficacy of the two fluids in relation to reduction in concomitant drug utilization, duration of ventilator usage, length of stay in ICU as well as total duration of hospitalization and neurocognitive status upto a period of 1 year post-CABG.

DETAILED DESCRIPTION:
Details provided in summary.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 45 to 80 years
* CABG patients with on or off pump procedure
* Ejection fraction < 50%
* Given informed consent

Exclusion Criteria:

* Combined operations
* Severe arrhythmia(VT, AF rapid response, heart blocks) and severe hemodynamic imbalance
* Severe bleeding and/or re-operation
* Hypernatremia > 155 mMol/L
* Severe liver failure(SGOT, SGPT 2x normal)
* Severe renal failure(Creatinine > 2 mg. %)
* Major diseases(eg. cancer)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hemodynamic status | During and 12 hours after CABG surgery

SECONDARY OUTCOMES:
Safety of hypertonic sodium lactate for maintaining hemodynamic stability | During and 12 hours after CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Leverve, MD, PhD, Principal Investigator — Director, INSERM-E0221-Bioenergetique Fondamentale et appliquee, Universite Joseph Fourier, France
Locations (1):
- National Cardiac Center, Department of Surgery and Intensive Care Unit, Harapan Kita Hospital, Jakarta, Jakarta Special Capital Region, Indonesia